CLINICAL TRIAL: NCT05184426
Title: MuLtimodality EvaluatiOn of aNtibody mEdiated Damage in Heart Transplantation (LEONE-HT)
Acronym: LEONE-HT
Status: Active, not recruiting | Type: Observational
Sponsor: Juan Francisco Delgado Jimenez (Other)
Collaborators: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor-Investigator, Juan Francisco Delgado Jimenez, Medical Director of Heart Transplant programme MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: LEONE-HT
Record Dates: First submitted 2021-07-19; First posted 2022-01-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Transplant Failure; Heart Transplant Rejection; Antibody-mediated Rejection
Keywords: Heart transplant; Anti-HLA antibodies; Magnetic Resonance; Echocardiogram; Transmission electron microscope
MeSH Terms: interventions — Echocardiography; Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endomyocardial biopsy samples Blood samples (leukocytes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Positive anti-HLA antibodies: Heart transplant patients who have developed antiHLA antibodies after transplant
  Interventions: Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Coronary angiography; Diagnostic Test: Endomyocardial biopsy
- Non-exposed: Negative anti-HLA antibodies: Heart transplant patients without antiHLA antibodies with similar transplant date to its correspondent case.
  Interventions: Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Coronary angiography; Diagnostic Test: Endomyocardial biopsy

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Ultrasound study to assess cardiac anatomy and function
Diagnostic Test: Cardiac magnetic resonance — MR to assess cardiac anatomy, function and tissue damage
Diagnostic Test: Coronary angiography — Cathteterization to assess coronary anatomy. Intravascular ultrasound to obtained a detailed assessment of vessels anatomy. Guidewire pressure to assess microcirculation
Diagnostic Test: Endomyocardial biopsy — Optic microscopy, immunofluorescence, transmission electron microscopy

SUMMARY:
Cross-sectional evaluation of antibody mediated injury in heart transplantation patients through a multimodal approach: electron microscopy, optic microscopy, immunohistochemistry techniques, transthoracic echocardiography, cardiac magnetic resonance, pressure guide wire, intravascular ultrasound

DETAILED DESCRIPTION:
Heart transplant survival has barely improved in the last decades and unsatisfactory for a large proportion of heart transplant recipients. The development of leukocyte antigen antibodies (anti-HLA) in the post-transplant patient is associated to the main causes of graft dysfunction. The mechanisms of this damage are unclear and there's no effective treatment.

The investigators aim is to identify early markers of graft injury through a complete morphological and functional evaluation with histological analysis, immunological assays, advanced imaging techniques and invasive evaluation of coronary vasculature in patients with anti-HLA compared to matching controls.

The investigators propose a cross-sectional study within a large heart transplant cohort. This is a multicentric observational multimodal study. The investigators aim is to establish early characteristics of antibody mediated damage and set the bases for future studies looking for new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

1. Exposed:

   * Heart transplant recipients
   * "De novo" antiHLA detection (after heart transplant):

     * Mean fluorescence intensity (MFI)) > 2000 for donor-specific antibodies
     * Standard fluorescence intensity (SFI) > 150 000 for non-donor specific antibodies
   * Detailed immunological history:

     * Determination of anti-HLA antibodies before heart transplant.
     * Serial determination of anti-HLA antibodies during heart transplantation follow-up
   * Known HLA typing of the donor.
2. Non-exposed: Heart transplant procedure contemporary to the index case with negative anti-HLA antibodies.

Exclusion Criteria:

* Recipient of a second HT
* Multiple organ transplantation
* Unknown immunological history
* Recipients sensitized with anti-HLA antibodies against donor's HLA before the transplant
* CMR contrast will not be administered in patients with glomerular filtration rate < 30 ml/kg/1.73m2
* Patients with implanted cardiac devices or any other magnetic resonance non-compatible metallic prosthetic material will not undergo CMR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be conformed of heart transplant patients who are under follow-up at 3 hospitals of the Autonomous Region of Madrid (Spain). All the three hospitals are national referral center for heart transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Histology findings with transmission electron microscopy (TEM) | 14 days
  Detailed description of the antibodies-mediated graft injury depending on exposition-time through a detailed evaluation
Histology findings with optic microscopy (OM) | 14 days
  Detailed description of the antibodies-mediated graft injury depending on exposition-time through a detailed evaluation
Histology findings with immunohistochemistry (IHQ) techniques. | 14 days
  Detailed description of the antibodies-mediated graft injury depending on exposition-time through a detailed evaluation

SECONDARY OUTCOMES:
Microvascular function (pressure guidewire) | 14 days
  Index of microcirculatory resistance
Microvascular function (pressure guidewire 2) | 14 days
  Coronary flow reserve
Microvascular function (cardiac magnetic resonance) | 14 days
  Quantitative perfusion evaluation
Increased water content (intracellular edema) | 14 days
  T2 recovery times mapping (cardiac magnetic resonance) to detect intracellular edema (endothelial vacuolization) as an early sign of microvascular damage
Myocardial fibrosis (cardiac magnetic resonance) | 14 days
  T1 recovery time mapping to identify remodeling and fibrosis secondary to microvascular damage
Myocardial fibrosis (cardiac magnetic resonance 2) | 14 days
  Extracellular volumen quantification to identify remodeling and fibrosis secondary to microvascular damage
Myocardial fibrosis (echocardiography) | 14 days
  Global longitudinal strain to identify remodeling and fibrosis secondary to microvascular damage
Serum markers of fibrosis | 14 days
  FGF - 23, PICP, PIIINP, galectin-3, soluble-ST2 as serum/plasmatic markers of fibrosis and remodeling
Coronary allograft vasculopathy (CAV) | 14 days
  Fractional flow reserve (coronary physiology) as early marker of CAV
Coronary allograft vasculopathy (CAV 2) | 14 days
  Intimal thickness (intravascular ultrasound) as early marker of CAV

OTHER OUTCOMES:
Adverse events | 5 years
  Heart failure, re-transplant, death

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Delgado, MD PhD, Study Chair — University Hospital 12 de Octubre
Locations (3):
- Spain (3):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nuche J, de la Cruz Bertolo J, Marco Clement I, Sanchez VS, Sarnago Cebada F, Mancebo E, Enguita AB, Alonso-Riano M, Ruiz-Hurtado G, Lopez-Azor JC, Hernandez-Perez FJ, Castrodeza J, Sanchez Gonzalez J, Arribas Ynsaurriaga F, Garcia-Cosio Carmena MD, Delgado JF. Rationale and Protocol of the Multimodality Evaluation of Antibody-Mediated Injury in Heart Transplantation (LEONE-HT) Observational Cross-Sectional Study. Methods Protoc. 2022 Sep 25;5(5):75. doi: 10.3390/mps5050075. PMID 36287047